CLINICAL TRIAL: NCT00005531
Title: Genetic Epidemiology of Sarcoidosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5064; R01HL054306 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-08

CONDITIONS: Lung Diseases; Sarcoidosis
MeSH Terms: conditions — Lung Diseases; Sarcoidosis

SUMMARY:
To determine if hereditary susceptibility predisposes African Americans to sarcoidosis and to identify sarcoidosis susceptibility genes in African Americans.

DETAILED DESCRIPTION:
BACKGROUND:

Sarcoidosis is a multisystem, granulomatous inflammatory disease of unknown etiology. Hereditary susceptibility to sarcoidosis is suggested by reports of familial clustering and a higher prevalence in certain ethnic groups, particularly African-Americans. Over four hundred kindreds been reported in the medical literature and these investigators have recently described 101 families and shown that African Americans have a higher prevalence rate of familial sarcoidosis than Caucasians (19 percent vs. 5 percent). The reasons why sarcoidosis clusters in families or the role of genetic factors in this disease are not known.

DESIGN NARRATIVE:

The study was carried out in African American families ascertained through 400 African American sarcoidosis patients evaluated at the Henry Ford Health System. They were tested for association of sarcoidosis with markers for candidate genes using the affected family-based control method and tested for possible environmental risk factors and genetic mechanisms of disease transmission by performing a segregation analysis in African American families.

A strong association of one or more of the candidate genes with sarcoidosis or an indication of major gene segregation for the disease, provided the basis for future linkage studies. Investigating the hereditary susceptibility of sarcoidosis was best done in African Americans, because of the greater severity and occurrence of disease in this population. Once the reasons for familial aggregation of sarcoidosis are determined, the etiology of this disease will be better understood and it should be possible to design new approaches to prevention and treatment.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) recor

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-12; Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Iannuzzi — Case Western Reserve University

REFERENCES:
- [Background] Rybicki BA, Maliarik MJ, Bock CH, Elston RC, Baughman RP, Kimani AP, Sheffer RG, Chen KM, Major M, Popovich J Jr, Iannuzzi MC. The Blau syndrome gene is not a major risk factor for sarcoidosis. Sarcoidosis Vasc Diffuse Lung Dis. 1999 Sep;16(2):203-8. PMID 10560124
- [Background] Rybicki BA, Maliarik MJ, Malvitz E, Sheffer RG, Major M, Popovich J Jr, Iannuzzi MC. The influence of T cell receptor and cytokine genes on sarcoidosis susceptibility in African Americans. Hum Immunol. 1999 Sep;60(9):867-74. doi: 10.1016/s0198-8859(99)00050-6. PMID 10527395
- [Background] Maliarik MJ, Rybicki BA, Malvitz E, Sheffer RG, Major M, Popovich J Jr, Iannuzzi MC. Angiotensin-converting enzyme gene polymorphism and risk of sarcoidosis. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1566-70. doi: 10.1164/ajrccm.158.5.9804123. PMID 9817709
- [Background] Maliarik MJ, Chen KM, Sheffer RG, Rybicki BA, Major ML, Popovich J Jr, Iannuzzi MC. The natural resistance-associated macrophage protein gene in African Americans with sarcoidosis. Am J Respir Cell Mol Biol. 2000 Jun;22(6):672-5. doi: 10.1165/ajrcmb.22.6.3745. PMID 10837363
- [Background] Rybicki BA, Kirkey KL, Major M, Maliarik MJ, Popovich J Jr, Chase GA, Iannuzzi MC. Familial risk ratio of sarcoidosis in African-American sibs and parents. Am J Epidemiol. 2001 Jan 15;153(2):188-93. doi: 10.1093/aje/153.2.188. PMID 11159165
- [Background] Rybicki BA, Elston RC. The relationship between the sibling recurrence-risk ratio and genotype relative risk. Am J Hum Genet. 2000 Feb;66(2):593-604. doi: 10.1086/302778. PMID 10677319
- [Background] Rybicki BA, Maliarik MJ, Poisson LM, Sheffer R, Chen KM, Major M, Chase GA, Iannuzzi MC. The major histocompatibility complex gene region and sarcoidosis susceptibility in African Americans. Am J Respir Crit Care Med. 2003 Feb 1;167(3):444-9. doi: 10.1164/rccm.2112060. PMID 12554629
- [Background] Rybicki BA, Iyengar SK, Harris T, Liptak R, Elston RC, Sheffer R, Chen KM, Major M, Maliarik MJ, Iannuzzi MC. The distribution of long range admixture linkage disequilibrium in an African-American population. Hum Hered. 2002;53(4):187-96. doi: 10.1159/000066193. PMID 12435883
- [Background] Kucera GP, Rybicki BA, Kirkey KL, Coon SW, Major ML, Maliarik MJ, Iannuzzi MC. Occupational risk factors for sarcoidosis in African-American siblings. Chest. 2003 May;123(5):1527-35. doi: 10.1378/chest.123.5.1527. PMID 12740270
- [Background] Iannuzzi MC, Maliarik MJ, Poisson LM, Rybicki BA. Sarcoidosis susceptibility and resistance HLA-DQB1 alleles in African Americans. Am J Respir Crit Care Med. 2003 May 1;167(9):1225-31. doi: 10.1164/rccm.200209-1097OC. Epub 2003 Feb 13. PMID 12615619